CLINICAL TRIAL: NCT06354348
Title: Practical Ultrasonographic Detection of Sarcopenia in Patients With Long-term Gastrectomy: A Cross-sectional Case-control Study
Brief Title: Practical Ultrasonographic Detection of Sarcopenia in Patients With Long-term Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Semih Sezer, clinic physician, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GastrectomyUSG
Record Dates: First submitted 2024-03-30; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Sarcopenia; Gastrectomy
MeSH Terms: conditions — Sarcopenia | interventions — Hand Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Total gastrectomy (Experimental): Patients with esophagojejunostomy on endoscopic evaluation were considered as total gastrectomy.
  Interventions: Diagnostic Test: USG, Grip strength, Chair stand test (CST)
- Distal gastrectomy (Experimental): Patients with resected mid-corpus with preserved corpus, fundus and cardia and gastrojejunostomy were considered as distal gastrectomy.
  Interventions: Diagnostic Test: USG, Grip strength, Chair stand test (CST)
- No gastrectomy status (Experimental): Has not undergone a gastrectomy operation
  Interventions: Diagnostic Test: USG, Grip strength, Chair stand test (CST)

INTERVENTIONS:
Diagnostic Test: USG, Grip strength, Chair stand test (CST) — Anterior thigh muscle thickness was measured with USG Grip strength was measured with an electronic hand dynamometer Chair stand test (CST) was performed while participants were asked to stand up and sit down from a chair - without arm rest, for five times as quick as possible, with their arms crossed over their chests.

SUMMARY:
The investigators aimed to evaluate long-term sarcopenia in patients with total and distal gastrectomy by measuring the anterior thigh muscle with USG, which is a more specific and easy method.

DETAILED DESCRIPTION:
Sarcopenia was found to be significantly increased in patients who underwent total, proximal and distal gastrectomy compared to those who did not undergo gastrectomy in the long term.

To date, very few studies have investigated the development of sarcopenia in the long term after gastrectomy. In these studies, sarcopenia was usually assessed using BIA and DEXA. Muscle thickness measured by ultrasound has high sensitivity and specificity in determining regional muscle mass.

Patients who underwent total(n=20) and subtotal gastrectomy(n=35) and patients who did not undergo gastrectomy(n=35) were included in the study.

Ultrasonographic measurements Anterior thigh muscle thickness of the dominant side was measured at the mid-point between the anterior superior iliac spine and the upper border of the patella. Transverse measurements were obtained between the outer fascia of rectus femoris muscle and the periosteum of femur. Sonographic thigh adjustment ratio (STAR) was calculated by dividing the anterior thigh muscle thickness (mm) by BMI.

Functional evaluations Grip strength was measured with an electronic hand dynamometer. Three repeat measurements were performed from the dominant side and the maximum value was taken for the analyses. Chair stand test (CST) was performed while participants were asked to stand up and sit down from a chair - without arm rest, for five times as quick as possible, with their arms crossed over their chests. Three measurements were performed and median values were taken for the analyses.

Diagnosis of sarcopenia The ISarcoPRM algorithm was used whereby the diagnosis of sarcopenia was established if low muscle mass (i.e. STAR values <1.4 for males and <1.0 for females) was combined with low grip strength (<32 kg (males) and <19 kg (females)) and/or increased CST time (≥12 sec).

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the study
* Total or subtotal gastrectomy at least 1 year ago
* The control group consisted of patients without gastrectomy with similar exclusion criteria as the patient group

Exclusion Criteria:

* Rheumatic/neurological diseases
* Any organ failure,
* Limitation of mobility
* History of major orthopedic surgery,
* Chemotherapy programs
* Gastric carcinoma recurrence
* Parkinson's disease, previous stroke, cerebellar diseases, multiple sclerosis
* Major depression
* Those who use any assistive device for walking
* People with severe knee, hip and hand osteoarthritis
* Active malignancies (currently or within the last 1 year receiving radiotherapy/chemotherapy
* Severe chronic obstructive pulmonary disease
* Visual impairment and vestibular disorders
* Pregnancy

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Sarcopenia (Sonographic thigh adjustment ratio (STAR) was calculated by dividing the anterior thigh muscle thickness (mm) by BMI ) | through study completion, an average of 4 months
  The diagnosis of sarcopenia was established if low muscle mass (i.e. STAR values <1.4 for males and <1.0 for females) was combined with low grip strength (<32 kg (males) and <19 kg (females)) and/or increased CST time (≥12 sec)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Kara M, Kaymak B, Frontera W, Ata AM, Ricci V, Ekiz T, Chang KV, Han DS, Michail X, Quittan M, Lim JY, Bean JF, Franchignoni F, Ozcakar L. Diagnosing sarcopenia: Functional perspectives and a new algorithm from the ISarcoPRM. J Rehabil Med. 2021 Jun 21;53(6):jrm00209. doi: 10.2340/16501977-2851. PMID 34121127
- [Background] Takahashi S, Shimizu S, Nagai S, Watanabe H, Nishitani Y, Kurisu Y. Characteristics of sarcopenia after distal gastrectomy in elderly patients. PLoS One. 2019 Sep 11;14(9):e0222412. doi: 10.1371/journal.pone.0222412. eCollection 2019. PMID 31509590
- [Background] Okamoto A, Aikou S, Iwata R, Oya S, Kawasaki K, Okumura Y, Yagi K, Yamashita H, Nomura S, Seto Y. The type of gastrectomy affects skeletal muscle loss and the long-term outcomes of elderly patients with gastric cancer: a retrospective study using computed tomography images. Surg Today. 2022 May;52(5):812-821. doi: 10.1007/s00595-021-02414-2. Epub 2021 Nov 26. PMID 34837102
- [Background] Kara M, Kaymak B, Ata AM, Ozkal O, Kara O, Baki A, Sengul Aycicek G, Topuz S, Karahan S, Soylu AR, Cakir B, Halil M, Ozcakar L. STAR-Sonographic Thigh Adjustment Ratio: A Golden Formula for the Diagnosis of Sarcopenia. Am J Phys Med Rehabil. 2020 Oct;99(10):902-908. doi: 10.1097/PHM.0000000000001439. PMID 32941253